CLINICAL TRIAL: NCT02889211
Title: Brain Function in Depression and Insulin Resistance
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Principal Investigator Left University
Sponsor: University of Pittsburgh (Other)
Responsible Party: Principal Investigator, John Patrick Ryan, Assistant Professor, University of Pittsburgh
Allocation: Non-Randomized | Model: Parallel | Masking: Single | Purpose: Basic Science
Other Study IDs: 16060315
Record Dates: First submitted 2016-08-23; First posted 2016-09-05 (Estimated); Last update posted 2017-12-05 (Actual); Status verified 2017-12

CONDITIONS: Depression; Insulin Resistance
MeSH Terms: conditions — Depression; Insulin Resistance

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No

ARMS (4):
- Metabolically Healthy - Non-depressed (Active Comparator): Overweight individuals without metabolic syndrome and free of psychiatric illness
  Interventions: Behavioral: Gambling Task
- Metabolically Healthy - Depressed (Experimental): Overweight individuals without metabolic syndrome and with active major depression
  Interventions: Behavioral: Gambling Task
- Insulin Resistant - Depressed (Experimental): Overweight individuals with metabolic syndrome and active major depression
  Interventions: Behavioral: Gambling Task
- Insulin Resistant - Non-depressed (Experimental): Overweight individuals with metabolic syndrome and free of psychiatric illness
  Interventions: Behavioral: Gambling Task

INTERVENTIONS:
Behavioral: Gambling Task

SUMMARY:
The purpose of this study is to help researchers learn about how the brain responds to rewards. This study is interested in seeing how these responses differ between people who are more and less responsive to insulin in their body, and people with and without depression.

ELIGIBILITY:
Inclusion Criteria:

Body Mass Index 24-34.9

HEALTHY CONTROLS HOMA-IR (fasting (glucose x insulin)/405) < 1.8

Not more than one of the following:

* Waist circumference > 40 inches (men) or > 35 inches (women)
* Triglycerides > 150 mg/dL
* HDL < 40 mg/dL (men) or < 50 mg/dL (women)
* Blood pressure > 135/85
* Fasting glucose > 100 mg/dL

INSULIN RESISTANT HOMA-IR > 2.0

And at least three of the following:

* Waist circumference > 40 inches (men) or >35 inches (women)
* Triglycerides > 150 mg/dL
* HDL < 40 mg/dL (men) or <50 mg/dL (women)
* Blood pressure > 135/85
* Fasting glucose > 100 mg/dL

MAJOR DEPRESSION, METABOLICALLY HEALTHY Meets criteria for MDD during SCID-5 evaluation HOMA-IR < 1.8

Not more than one of the following:

* Waist circumference > 40 inches (men) or >35 inches (women)
* Triglycerides > 150 mg/dL
* HDL < 40 mg/dL (men) or <50 mg/dL (women)
* Blood pressure > 135/85
* Fasting glucose > 100 mg/dL

MAJOR DEPRESSION, INSULIN RESISTANT Meets criteria for MDD during SCID-5 evaluation HOMA-IR > 2.0

And at least three of the following:

* Waist circumference > 40 inches (men) or >35 inches (women)
* Triglycerides > 150 mg/dL
* HDL < 40 mg/dL (men) or <50 mg/dL (women)
* Blood pressure > 135/85
* Fasting glucose > 100 mg/dL

Exclusion Criteria:

* - History of mania or psychosis
* Current suicidal ideation
* Alcohol or substance abuse including cannabis use (current or in the last three months)
* Early onset dementia of any etiology
* Medical conditions with known significant effects on mood (e.g. Stroke or current hypothyroid state)
* Unstable medical illnesses (e.g. Delirium, uncontrolled DM, uncontrolled cardiovascular illness)
* Use of high doses of benzodiazepines (> 2mg lorazepam/day equivalent)
* Given the high comorbidity (80%) between MDD and anxiety disorders, participants with comorbid anxiety disorders will be included in the study as long as the clinical presentation suggests that depression precedes the onset of anxiety
* Current or lifetime history of cancer, a chronic kidney or liver condition, type I or II diabetes
* Current or lifetime use of glucocorticoid medications for >1 month
* Previous cerebrovascular accident or trauma involving loss of consciousness
* Previous neurosurgery or history of a neurological condition
* Pregnancy (females)
* Claustrophobia
* Ferrous metallic implants or any surgically placed medical device not cleared for safety at 3Tesla MRI strength
* Positive Hepatitis C serology or other known viral infections that may induce insulin resistance
* Peripheral vascular disease
* Liver, kidney, or active blood disease
* Peripheral neuropathy
* Fasting glucose > 126 mg/dL
* Currently taking any medications that can alter glucose homeostasis (steroids, glucocorticoids, nicotinic acid)
* Currently taking thiazolidinediones or insulin
* Females currently on hormone replacement therapy (HRT) less than 6 months
* Being left handed
* Use of antidepressant medication within the past two weeks (six weeks fluoxetine)
* Suicide risk
* Current use of stimulants, antipsychotic medications, mood stabilizers, cognitive enhancers, statins, glucocorticoids, steroids, nicotinic acid, thiazolidinediones, insulin, metformin, any diabetes medications (e.g. gliptins), HIV medications.

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 42 (Actual)
Dates: Start 2016-08; Primary Completion 2017-12 (Actual); Study Completion 2017-12 (Actual)

PRIMARY OUTCOMES:
fMRI BOLD Response in Striatal Regions | During Gambling Task in fMRI Scanner
  The investigators will monitor the blood oxygen level dependent response using fMRI and compare activation during "win" trials vs. "loss" trials

CONTACTS AND LOCATIONS:
Locations (1):
- Western Psychiatric Institute and Clinic at University of Pittsburgh, Pittsburgh, Pennsylvania, United States

IPD SHARING:
Plan to Share IPD: No